CLINICAL TRIAL: NCT03476291
Title: Research of Automated Maculopathy Screening by Optical Coherent Tomography Image-based Deep Learning Techniques
Brief Title: Research of Automated Maculopathy Screening Based on AI Techniques Using OCT Images
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: JSPH-AIOCT-001
Record Dates: First submitted 2018-02-26; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-02

CONDITIONS: Maculopathy
Keywords: macular diseases; screening; OCT; Deep learning; AI
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal: normal macular structure of horizontal OCT B-scans
- Abnormal: abnormal macular structure of horizontal OCT B-scans, including many sub-categories of pathological features, like epiretinal membrane, pigment epithelium detachment, ect.

SUMMARY:
The investigators expect to develop an algorithm that can interpret OCT images and automated determine whether the macula is normal or not by using OCT image-based deep learning techniques. And investigators wish to develop software applications that will help better screen and diagnose macular diseases in resource-limited areas.

DETAILED DESCRIPTION:
The investigators will apply deep learning convolutional neural network by using ImageNet for an automated detection of multiple retinal diseases with OCT horizontal B-scans with a high-quality labeled database. Datasets, including training dataset, testing dataset and validation datasets, will be built by ophthalmologists of the First affiliated hospital of Nanjing Medical University according to the standardized annotation guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending the Ophthalmology Department of the First Affiliated Hospital of Nanjing Medical University within 5 years and who received known, clear diagnoses with digital retinal imaging (including OCT, fundus digital photographs and fundus fluorescein angiography, at least with OCT images) as part of their routine clinical care, will be eligible for inclusion in this study.

Exclusion Criteria:

* Hardcopy examinations (i.e., photos of paper reports of OCT imaging performed at other hospitals) will be ineligible.
* Data from patients who have previously manually requested that their data should not be shared, even for research purposes in anonymised form, and have informed the Ophthalmology Department of the First Affiliated Hospital of Nanjing Medical University of this desire (even in previously conducted studies or other on-going studies in this hospital), will be excluded, and their data will not be upload to the cloud platform before research begins.
* Data from eyes tamponed with silicone oil or gas (i.e., C3F8) will be ineligible.
* Data with poor image quality, such as incomplete images, inverted images, blurred or cracked images and images with a very weak signal (i.e., vitreous haemorrhage), will be ineligible.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: no age limited, no gender-based
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
receiver operating characteristic(ROC) curve of the algorithm | approximately 1 year
  It is also called sensitivity curve. The ROC curve shows how sensitive the algorithm model is to automatically detect the desired output.
Area under the ROC curve(AUC) | approximately 1 year
  It shows the operating value of the algorithm model, which can represent the effect of the model.

CONTACTS AND LOCATIONS:
Overall Officials: Songtao Yuan, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No